CLINICAL TRIAL: NCT06870409
Title: A Prospective Interventional Randomized Placebo-controlled Multicenter Clinical Trial of the Efficacy, Tolerability and Safety of Phage Therapy in Combination With Standard Antibiotic Therapy in Patients With Infective Endocarditis
Brief Title: Bacteriophages in Addition to Antibiotics for the Treatment of Patients With Infective Endocarditis
Acronym: PHARAOH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Clinical Hospital na V.V.Vinogradov (branch of RUDN university na Patrice Lumumba) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BP-IE-2024
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Endocarditis, Bacterial
Keywords: infective endocarditis; bacteriophages
MeSH Terms: conditions — Endocarditis, Bacterial; Endocarditis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Patients with infective endocarditis will receive a placebo in addition to standard antibiotic therapy
  Interventions: Drug: Bacteriophage
- Bacteriophage (Experimental): Group of patients who will be supplemented with bacteriophage complex drug in addition to standard antibiotic therapy
  Interventions: Drug: Bacteriophage

INTERVENTIONS:
Drug: Bacteriophage — Complex drug of 3-4 virulent phages to each type of bacteria, active against:
  * Staphylococcus spp. [Staphylococcus aureus, CoNS (S. epidermidis, S. haemolyticus, S. hominis, S. warneri, S. capitis)].
  * Streptococcus spp. [Streptococcus viridans (Str. mutans, Str. sanguis, Str. mitis, Str. cristatus, Str. gordonii, Str. oralis, Str. salivarius), Gemella hemolysans, Str. bovis (Str. gallolyticus), Str. constellatus, Str. anginosus, Str. agalactiae].
  * Enterococcus spp. [E. faecalis, E. faecium].
  * Non-HACEK [E. coli, A. baumanii, K. pneumoniae, P. aeruginosa]

SUMMARY:
Infective endocarditis (IE) is an endocardial lesion caused by bacterial and/or fungal infection that most commonly affects the heart valves and/or the endocardium around implanted intracardiac devices. In general, IE is classified as a rare disease, but there has been a steady increase in incidence, primarily in high-income countries. The danger of IE lies in the high frequency of complicated course of the disease and the risk of lethal outcomes both at the inpatient stage of treatment 25.0% and in the distant period 30-40%. The annual incidence is from 3 to 10 per 100,000 people.

In addition to the difficulties in the diagnosis of IE, the most challenging aspect is the prescription of effective antibiotic therapy, especially in the context of unidentified etiology of IE and the growth of multi-resistant pathogens. Many solutions are used to achieve successful therapy of IE, including the prescription of combined antibiotic therapy, the use of new modern antibacterial drugs, the prescription of therapy taking into account the sensitivity of the pathogen, but the failure of treatment and the number of resistant pathogens are only increasing. Moreover, antibacterial therapy is relevant both in patients on conservative treatment of IE and after cardiac surgery, among whom the risk of nosocomial or healthcare-associated infections is additionally increased. Thus, new ways of modernising IE therapy are needed. Phage therapy is considered one of the promising strategies [6-8]. Bacteriophages are certain viruses that naturally infect bacteria and are used as antibacterial treatments. Phagotherapy is used as antibacterial drugs that can induce lysis of target pathogens.

DETAILED DESCRIPTION:
Given the steady increase in antibiotic resistance in bacteria and the decreasing number of new antibacterial drugs, phage therapy may prove to be a revolutionary safe approach, especially attractive for the following reasons: phages are easily isolated from a diverse environment and affect only the pathogenic cell without affecting neighbouring cells, they are able to successfully target bacteria with multiple resistance and, therefore, can potentially replace antibiotic therapy. A feature of bacteriophages is their high specificity, which at the same time may be a limitation for their widespread use in the absence of knowledge about bacterial sensitivity. The above-mentioned suggests the possibility of using a cocktail of bacteriophages selected taking into account the expected spectrum of pathogens and their sensitivity. A similar strategy was first developed by Zurabov F. (2021), who proposed adaptive phagotherapy for the prevention of recurrent nosocomial pneumonia, the specificity of which was the selection of bacteriophages not for an individual patient, but for the entire spectrum of bacteria circulating in the intensive care unit with continuous clinical and microbiological studies with monitoring of efficacy. Based on the collection of hospital bacteria of 66 antibiotic-resistant strains, a complex preparation of bacteriophages for inhalation administration was developed. The study included 83 patients in chronic critical condition with recurrent pneumonia in whom high safety and efficacy of the new approach were convincingly demonstrated. The undeniable advantage of phagotherapy is its targeted effect on pathogenic bacteria without affecting the microbiota, and therefore the absence of such side effects as mucous membrane candidiasis, antibiotic-associated diarrhoea, pseudomembranous colitis, etc. A number of studies have demonstrated the absence of any side effects, which is probably due to the fact that bacteriophages are natural inhabitants of the environment in harmony with humans. A number of studies have demonstrated the absence of any side effects, which is probably due to the fact that bacteriophages are natural inhabitants of the environment, harmoniously co-existing with humans. A separate advantage of phage therapy is the ability of several types of phages to affect the same bacterial strains, which minimises the risk of developing resistance to bacteriophages.

The success of phagotherapy in patients with IE has been demonstrated in only a small number of experimental and clinical studies. The treatment with BF does not yet have a strong evidence base from randomised clinical trials, but the available clinical data from a variety of pathologies (skin, soft tissue and joint infections, implanted intracardiac devices), suggest that phage therapy may be an effective adjunct to conventional antibiotic therapy or even as a stand-alone treatment.

Since currently the most common pathogens of IE are staphylococci, in particular S. aureus, the largest number of studies on the use of BF has been noted in this etiological affiliation of IE. As S. aureus-induced IE is more often associated with an unfavourable course, this is what prompted the search for new approaches to therapy, and the first studies on the use of BF represented a salvage therapy, especially in the context of multidrug resistance. In general, no more than 10 modern experimental and clinical studies on the possibility of using bacteriophages in staphylococcal IE are presented, including 3 separate clinical observations and one description of a series of 13 cases of IE. In an experimental rat model of S. aureus MSSA IE showed high efficacy of combined therapy with flucloxacillin with phage cocktail (intravenous form) with respect to vegetation sterility in 9/12 rats. Similar success was obtained in the experiment of IE caused by S. aureus MRSA when treated with a combination of bacteriophages with vancomycin. This type of pathogen is characterised by a high incidence of antibiotic resistance, which makes the use of BF in this group of patients particularly useful. In 2019 was one of the first to present a clinical observation of a 65-year-old patient with non-ischaemic dilated cardiomyopathy and IE of intracardiac device, uncontrolled course of infection against the background of repeated change of antibiotic therapy. The use of intravenous anti-staphylococcal cocktail AB-SA01 for 28 days 2 times a day in combination with antibiotic therapy allowed to achieve complete control of infection with subsequent heart transplantation [30]. In 2019 was demonstrated a similar observation of successful application of intravenous anti-staphylococcal cocktail AB-SA01 for 14 days twice a day in a patient with IE of S. aureus prosthetic valve and ineffectiveness of antibiotic therapy. Combined treatment with BF allowed to achieve complete recovery of the patient. The efficacy and safety of intravenous anti-staphylococcal cocktail AB-SA01 for 14 days twice a day in 13 patients with severe S.aureus infections, including IE. The researchers did not note any side effects, but the conclusion on the efficacy of therapy required further studies.

Pneumococcal bacteriophage Cpl-1 was investigated in an experiment on rats with IE caused by Str. pneumoniae, demonstrating rapid blood sanitation and reduction of pathogen concentration in vegetations. Also, researchers investigated the efficacy of phage therapy in IE caused by Pseudomonas aeruginosa in an experiment. The combination of BF and ciprofloxacin caused rapid sanitation of vegetations.

Among the dangerous and difficult to treat pathogens of IE, it is necessary to highlight the representatives of enterococci - Ent. faecalis and Ent. faecium, characterised by the ability to develop multidrug resistance, which has increased markedly over the last 10 years. According to some data, the incidence of enterococci in fatal IE can reach 97%. A distinctive feature of enterococci is their ability to form biofilms, which significantly complicates the therapy of IE. BF has a unique ability to destroy biofilms based on the layer-by-layer penetration of BF into deeper layers of vegetation. In an experiment proved that BFs are able to penetrate vegetations, including in IE caused by E. faecalis. There have been no clinical studies on the efficacy of BF in enterococcal IE. In an experiment on modelling vegetations from human blood ex vivo, another study showed the possibility of synergy of BF with antibacterial drugs (daptomycin, ceftraroline), including the restoration of sensitivity of enterococci to antibacterial drugs.

Thus, the treatment of IE, even with a known etiology, is a global challenge. Considering the fact that IE is often found among comorbid, elderly and debilitated patients, with high cardiac surgery perioperative risk, as well as the high frequency of IE with unidentified etiology not because of association with hard-to-cultivate pathogens, but because of low concentration of typical pathogen in blood due to previous antibiotic therapy, prolonged effective antibiotic therapy is often the only safe solution in such cases. Taking into account the limited spectrum of effective antibacterial drugs, it is extremely important to study the efficacy and safety of phagotherapy in combination with antibacterial drugs in IE. The most optimal is the study of phagotherapy in the form of phage cocktail to the most common typical pathogens of IE with application at the initial stages of treatment as part of empirical antibacterial therapy. It is assumed that such an early start of effective treatment will avoid the development of resistance to antibacterial drugs and lead to rapid relief of IE activity with subsequent transfer of patients to outpatient treatment regimes. The advantage of the presented treatment algorithm is the possibility to cover all patients with IE before the etiological affiliation is established, which will make it possible to obtain the treatment effect already at the early stages of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation with active IE or active IE developed in hospital;
* Definite diagnosis of IE according to modified Duke 2023 criteria or possible diagnosis of IE but managed and treated as IE;
* Informed consent to participate in the study;

Exclusion Criteria:

* Inactive (transferred) IE
* Non-bacterial thrombotic endocarditis
* Active oncological diseases
* Immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2028-02-05 (Estimated); Study Completion 2029-02-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of the combined endpoint (duration of hospitalisation > 14 days , hospital embolic events and death) in patients with IE receiving adjunctive therapy with bacteriophage complex preparation in combination with standard antibiotic therapy | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Hospital named after V.V.Vinogradov (branch) of the Peoples' Friendship University of Russia named after Patrice Lumumba, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: unlimited
Access Criteria: anyone